CLINICAL TRIAL: NCT06436378
Title: Feasibility and Efficacy of Music Intervention on Pain, Anxiety, and Well-being in Chronic Pain Patients
Brief Title: Music Intervention in Chronic Pain Patients
Acronym: MusicCPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Principal Investigator, Josiane Bissonnette, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-6620
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Chronic Pain; Anxiety; Well-Being, Psychological
Keywords: chronic pain; music; anxiety; well-being
MeSH Terms: conditions — Chronic Pain; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Musical intervention (Experimental): This arm will receive a personalized music intervention.
  Interventions: Behavioral: Music intervention in person
- No musical intervention (No Intervention): This arm will carry out its daily activities and will be assessed using the same measures at the beginning of each session and after a delay comparable to the duration of the intervention administered in the experimental group.

INTERVENTIONS:
Behavioral: Music intervention in person — The music intervention consists of listening to two or three pieces of music chosen by each participant that bring them a sense of well-being. One of the two music intervention sessions will be preceded by a moment of relaxation, during which participants will be asked to focus their attention on their breathing, on relaxation, and on the process of self-absorption. This intervention, preceded by a brief moment of relaxation, will take place during the first session for half of the participants and during the second session for the other half.
  Arms: Musical intervention

SUMMARY:
The goal of this randomized controlled trial is to evaluate the efficacy of a personalized music intervention program to improve the condition of individuals suffering from chronic pain.

The main objective is to evaluate if the intervention program will significantly reduce participants composite score of pain, anxiety, and well-being (reversed) as evaluated by the Edmonton symptom assessment scale (ESAS-r) immediately after the intervention, and whether this improvement will be significantly greater than that of control sessions.

DETAILED DESCRIPTION:
The participants (n = 36) will be randomized into two groups. The intervention will last for 4 weeks. Once per week for the first 2 weeks, the first group will have a personalized musical intervention in person on the university campus and will evaluate their pain, anxiety, and well-being scores before and after each session. For the following 2 weeks, the participants will have online access to their music sessions and will also assess their levels of pain, anxiety, and well-being before and after each intervention session.

The second group (control group) will evaluate their pain, anxiety, and well-being scores 20 minutes apart once per week for the first 2 weeks.Participants will continue their daily activities between the two measurement times. During the next 2 weeks, the participants will listen to online musical sessions once per week and will again evaluate their levels of pain, anxiety, and well-being before and after each intervention session.

The main objective of this randomized controlled trial is to evaluate the immediate effect of a personalized music intervention for the experimental group/in-person intervention on a composite score of pain, anxiety, and well-being (reversed), compared to the control group/no intervention sessions, as measured by the ESAS-r. The secondary objective is to assess the evolution of each of these three ESAS-r variables (pain, anxiety, well-being) from pre-test to post-test compared with changes in these variables in the control group/no intervention sessions.

The differences between in-person musical interventions and online musical sessions, as well as the feasibility and adherence of participants to an online music intervention program, will also be assessed. Furthermore, the effect of a music session preceded by a period of relaxation compared to the effect of a musical session alone, and the experiential dimensions experienced, will be evaluated.

At the end of the experiment, both groups will be interviewed to analyze their comments regarding the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older;
* Suffering from chronic pain and actively attending the pain clinic at the CHU de Québec-Université Laval;
* Have an email and be able to respond to online questionnaires using a computer, tablet, or phone;
* Have satisfactory or corrected hearing;
* Understand French;
* Be able to travel to Université Laval.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All
Enrollment: 36 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Composite pain, anxiety, and well-being (reversed) score | The posttest was administered 25 minutes after the pretest
  Change in composite outcome score for pre-test to post-test for the experimental sessions compared with change in the control sessions. The composite score will be obtained by summing the pain (0-10), anxiety (0-10) and well-being (reversed) scores (0-10) from the Edmonton Symptom Assessment Scale Revised. (ESAS-r)

SECONDARY OUTCOMES:
Changes in Pain levels | The posttest was administered 25 minutes after the pretest.
  Change in pain level, as assessed by the Edmonton Symptom Assesment Scale Revised (ESAS-r) on a scale of 0 to 10.
Changes in Anxiety levels | The posttest was administered 25 minutes after the pretest.
  Change in anxiety level, as assessed by the Edmonton Symptom Assesment Scale Revised (ESAS-r) on a scale of 0 to 10.
Changes in well-being (reversed) | The posttest was administered 25 minutes after the pretest.
  Change in well-being (reversed) level, as assessed by the Edmonton Symptom Assesment Scale Revised (ESAS-r) on a scale of 0 to 10.

OTHER OUTCOMES:
Subjective experience | 5 week
  Five open questions will be asked by the facilitator to inquire about the participant's experience. - Tell me about your experience with the intervention program. - What is your overall opinion of the intervention? - What did listening to the recordings bring you? - What did you like least about the intervention? - What would you change about the intervention? - Have you had any prior experience with this type of intervention?

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie Pinard, Md, MA, Principal Investigator — CIRRIS
Locations (1):
- Pavillon Louis-Jacques-Casault, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No